CLINICAL TRIAL: NCT01268748
Title: Efficacy of Transumbilical Versus Standard Laparoscopic Cholecystectomy on Postoperative Pain
Brief Title: Single Port Versus Four Ports Laparoscopic Cholecystectomy and Early Postoperative Pain
Acronym: UMBI-CHOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Lars Nannestad Jorgensen MD, DrMSc, Professor, Dept. of Surgery K, Bispebjerg Hospital, University of Copenhagen, DK-2400 Copenhagen NV, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-3-2010-064
Record Dates: First submitted 2010-09-20; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-09

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications
Keywords: single site surgery; laparoscopic surgery; pain; nausea
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications; Pain; Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 ports laparoscopic cholecystectomy (Other)
  Interventions: Procedure: Conventional laparoscopic procedure
- One port transumb. laparoscopic surgery (Other)
  Interventions: Procedure: Experimental laparoscopic procedure

INTERVENTIONS:
Procedure: Conventional laparoscopic procedure — Patients allocated to this group will undergo laparoscopic cholecystectomy using two 12 mm ports and two 5 mm ports
  Other Names: Versaport 12 mm; Versaport 5 mm
  Arms: 4 ports laparoscopic cholecystectomy
Procedure: Experimental laparoscopic procedure — Patients allocated to this group will undergo laparoscopic cholecystectomy using only a transumbilical SILS port
  Other Names: SILS port
  Arms: One port transumb. laparoscopic surgery

SUMMARY:
This is a trial to evaluate if single port laparoscopic cholecystectomy causes less pain than conventional laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This study is a randomized, two-arm, double-blinded three-center trial to compare single-port transumbilical laparoscopic cholecystectomy with conventional 4-port laparoscopic cholecystectomy. 120 patients are included with a 1:1 randomization. Three centers participate in the trial.

Inclusion criteria: Female patients, ASA I-III, age between 18 and 75 years, elective laparoscopic cholecystectomy because of biliary pain or recent uncomplicated biliary pancreatitis.

Exclusion criteria: Expected poor compliance, history of cholecystitis or severe pancreatitis, previous open upper abdominal surgery, pregnancy or lactation, preoperative chronic pain or conversion from laparoscopic to open surgery.

Pain and nausea is measured on VAS before the operation and 3 hrs, 1 day, 2 days and 3 days after the operation.

Cosmesis is evaluated after 28 days.

Patients are telephone-interviewed after 12 months and asked about port hernia formation. If hernia is suspected patients are called in for an abdominal ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Planned elective laparoscopic cholecystectomy because of biliary pain or uncomplicated biliary pancreatitis

Exclusion Criteria:

* Expected poor compliance
* History of cholecystitis or severe pancreatitis
* Earlier open upper abdominal surgery, pregnancy or lactation, chronic pain or conversion to open surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Pain scores on the Visual Analog Scale before surgery | Before surgery
Pain scores on the Visual Analog Scale 3 hours after surgery | 3 hrs after surgery
Pain scores on the Visual Analog Scale 1 day after surgery | 1 day after surgery
Pain scores on the Visual Analog Scale 2 days after surgery | 2 days after surgery
Pain scores on the Visual Analog Scale 3 days after surgery | 3 days after surgery

SECONDARY OUTCOMES:
Nausea scores on a 4 point scale before surgery | Before surgery
  The 4 point scale: none, light, moderate, and severe
Nausea scores on a 4 point scale 3 hours after surgery | 3 hours after surgery
  The 4 point scale: none, light, moderate, and severe
Nausea scores on a 4 point scale 1 day surgery | 1 day after surgery
  The 4 point scale: none, light, moderate, and severe
Nausea scores on a 4 point scale 2 days after surgery | 2 days after surgery
  The 4 point scale: none, light, moderate, and severe
Nausea scores on a 4 point scale 3 days after surgery | 3 days after surgery
  The 4 point scale: none, light, moderate, and severe
Well being scores on the Visual Analog Scale before surgery | Before surgery
Well being scores on the Visual Analog Scale 3 hours after surgery | 3 hours after surgery
Well being scores on the Visual Analog Scale 1 day after surgery | 1 day after surgery
Well being scores on the Visual Analog Scale 2 days after surgery | 2 days after surgery
Well being scores on the Visual Analog Scale 3 days after surgery | 3 days after surgery
Number of participants with adverse events as a measure of safety and tolerability | Within 30 days after surgery
  Adverse events include all complications related to surgery
Patient-assessed cosmesis on the Visual Analog Scale 30 days after surgery | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haytham Al-Tayar, MD, Principal Investigator — Dept. of Surgery, Bispebjerg Hospital, University of Copenhagen; Sami Assaadzadeh, MD, Principal Investigator — Dept. of Surgery, Gentofte Hospital, University of Copenhagen; Jacob Rosenberg, MD, DrMSc, Principal Investigator — Dept. of Surgery, Herlev Hospital, University of Copenhagen; Flemming Hjørne, MD, Principal Investigator — Dept. of Surgery, Køge Hospital, University of Copenhagen; Thue Bisgaard, MD, DrMSc, Principal Investigator — Dept. of Surgery, Køge Hospital, University of Copenhagen
Locations (3):
- Denmark (3):
  - Dept. of Surgery K, Bispebjerg Hospital, Copenhagen NV
  - Gentofte Hospital, University of Copenhagen, Gentofte Municipality
  - Dept. of Surgery, Koege Hospital, University of Copenhagen, Koege

REFERENCES:
- [Derived] Jorgensen LN, Rosenberg J, Al-Tayar H, Assaadzadeh S, Helgstrand F, Bisgaard T. Randomized clinical trial of single- versus multi-incision laparoscopic cholecystectomy. Br J Surg. 2014 Mar;101(4):347-55. doi: 10.1002/bjs.9393. PMID 24536008